CLINICAL TRIAL: NCT04984629
Title: Prospective, Single Arm, Non-randomized, Traditional Feasibility Study to Evaluate the Safety and Performance of the ReGelTec HYDRAFIL System
Brief Title: Study of the ReGelTec HYDRAFIL System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ReGelTec, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGOUS -1000CAN
Record Dates: First submitted 2021-07-14; First posted 2021-07-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Degenerative Disc Disease
Keywords: DDD; Degenerative Disc Disease; Back Pain; Lumbar Pain
MeSH Terms: conditions — Intervertebral Disc Degeneration; Back Pain; Low Back Pain

STUDY DESIGN:
Intervention Model Description: All subjects will receive the HYDRAFIL implant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HYDRAFIL Implant (Experimental): Polymer Implant of HYDRAFIL into a one or two lumbar intervertebral discs
  Interventions: Device: HYDRAFIL

INTERVENTIONS:
Device: HYDRAFIL — The HYDRAFIL System contains the following items: the Delivery System and the Pressure Gauge. The HYDRAFIL implant is contained within a pre-filled syringe that is inserted into the delivery system housing during the manufacturing process. The implant is heated within the delivery system prior to use to ensure a flowable implant that can be injected through a standard coaxial needle.

SUMMARY:
A study designed to treat patients with back pain associated with degenerative lumbar disc disease.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety and effectiveness of the ReGelTec HYDRAFIL System in subjects with axial low back pain (LBP) due to degenerative disc disease (DDD) who continue to have severe back pain and dysfunction after at least six (6) months of conservative care.

The primary objective of this study is to evaluate the safety and efficacy the HYDRAFIL System.

ELIGIBILITY:
Inclusion Criteria:

* Present with predominant low back pain and symptoms of DDD of the lumbar region of at least 6 months duration
* Failure to have their symptoms resolve or reduce following 6 months conservative care (pain medication and/or physical therapy)
* Male or female patients aged 22 to 80 years, inclusive
* Presence of DDD on magnetic resonance imaging (MRI) scan with global disc degeneration. Modified Pfirrmann grades 5 to 8 as characterized by MRI
* The presence of one or two symptomatic discs exhibiting degeneration contained within a competent outer annulus as determined by MRI and provocative discography and/or anaesthetic discography at L1-S1
* Patients who are legally competent and able to understand the nature, scope and aim of the clinical investigation
* Signed an informed subject consent form in a language in which they are fluent

Exclusion Criteria:

* History of or current systemic or local infection
* Annular tear or defect that shows free contrast extravasation into the epidural space during or after discography
* Presence of disc herniation that accounts for the majority of the patient's symptoms
* Subjects with Modic type 3 changes
* Subjects with trans-endplate disc herniations or Schmorl's nodes
* Neurogenic claudication due to spinal stenosis
* Previous back surgery at the target level of the lumbar spine
* Evidence of severe compression of cauda equina
* Spinal segmental instability (spondylolysis or spondylolisthesis: Grade >1), spinal canal stenosis, isthmus pathology, scoliosis [Cobb angle >20 at the incident level] and other deformity conditions that may compromise the study
* Subjects with arachnoiditis
* Subjects who are prisoners or wards of the courts
* Subjects involved in active litigation including worker's compensation cases
* Subjects with low back pain of non-spinal or unknown etiology
* Subjects with severe osteoporosis or metabolic bone disease
* Subjects who have a history of or are current abusers of alcohol or drugs (using definition criteria from the Diagnostic and Statistical Manual of Mental Disorders (DSM-V))
* If female, patients who are pregnant or are trying to become pregnant during the course of the trial. (due to risks of additional radiation exposures)
* Failure to understand informed consent or participation in any other clinical study
* Body Mass index (BMI) greater than 40
* Patients with active tumors in the spinal region
* Patients who have been diagnosed to diabetes mellitus
* Patients who have a sensitivity or allergy to the implant materials

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Success | post-treatment
  Successful implantation of the ReGelTec HYDRAFIL System implant in a lumbar disc nucleus

SECONDARY OUTCOMES:
Back pain as measured by NRS | 3, 6, 12 and 24 months
  Decrease in Numeric Rating Scale (NRS) Score - Back Pain
Function as measured by ODI | 3, 6, 12 and 24 months
  Maintenance of, or further improvement in the Oswestry Disability Index (ODI) Score
Safety of the ReGelTec Implant by demonstrating durability over the long term and no unanticipated safety concerns that arise | 3, 6, 12 and 24 months
  Freedom from Device or Operative Related Serious Adverse Events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Clerk-Lamalice, MD, MSc, FRCPC, FIPP, Principal Investigator — Beam Interventional & Diagnostic Imaging
Locations (1):
- Beam Interventional & Diagnostic Imaging, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor Website — http://www.regeltec.com